CLINICAL TRIAL: NCT03874416
Title: A Randomized Controlled Trial of Cognitive Rehabilitation of Working Memory After Moderate to Severe Traumatic Brain Injury
Brief Title: Cognitive Rehabilitation of Working Memory After Moderate to Severe Traumatic Brain Injury
Acronym: REHAB-MDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K160902J; PHRIP-16-0380 (Other: Ministry of health); 2018-A02713-52 (Registry Identifier: IDRCB (ANSM))
Record Dates: First submitted 2019-02-04; First posted 2019-03-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Moderate to Severe Traumatic Brain Injury
Keywords: moderate to severe traumatic brain injury; cognitive rehabilitation; working memory; daily life function; Working Memory Questionnaire, WMQ; Brown-Peterson test

STUDY DESIGN:
Intervention Model Description: Single blind trial with 2 parallel arms:
  Specific rehabilitation of working memory vs. non-specific rehabilitation
Who Masked: Outcomes Assessor
Masking Description: Clinical assessment will be performed by an assessor blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific rehabilitation of working memory (Experimental): Specific rehabilitation of working memory according to hierarchized rehabilitation.
  Interventions: Other: Specific rehabilitation
- Control group (Active Comparator): Non-specific rehabilitation of working memory, usual therapy.
  Interventions: Other: Non-specific rehabilitation

INTERVENTIONS:
Other: Specific rehabilitation — Experimental rehabilitation of working memory:
  3 sessions per week during 3 months, for a total 36 sessions.
  Arms: Specific rehabilitation of working memory
Other: Non-specific rehabilitation — Usual non-specific rehabilitation treatment for moderate to severe TBI in healthcare facilities: 2-3 sessions per week for 3 months.
  Arms: Control group

SUMMARY:
The study aims to demonstrate improvement of daily life functioning and improvement of cognitive tests in post traumatic brain injury (TBI) patients suffering from working memory deficit, by a 3-month specific cognitive rehabilitation program, in comparison with patients with usual non-specific rehabilitation of same duration.

As secondary objectives, the study aims to:

* demonstrate improvement of specific neuropsychological tests of working memory;
* demonstrate improvement of non-specific tasks involving working memory;
* assess the evolution in not-targeted domains by the specific rehabilitation, which would give evidence of a global cognitive stimulation effect;
* demonstrate improvement of social integration ability and quality of life;
* demonstrate persistence of effects at 3 months and 6 months after the end of treatment;
* demonstrate the acceptability, the tolerance and the feasibility of rehabilitation.

DETAILED DESCRIPTION:
Working memory is an essential cognitive function which allows to store briefly and treat simultaneous informations, but is often altered after a moderate to severe TBI. This alteration results in disabilities and social integration difficulties in the post TBI patients. The study team had developped a standardized and hierarchized rehabilitation program of working memory. Several experiments have shown the efficacy of the program which is now used in routine care by speech-language pathologists and neuropsychologists. However it is necessary to provide a robust demonstration of its efficacy in improving function in daily life.

This randomized multicenter study will be performed in 6 centers in the area of Île-de-France. 54 patients will be randomized 1:1 to receive either specific rehabilitation of working memory or non-specific rehabilitation. A 10-month follow-up is planned for patients of the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 - 65 years;
* Moderate to severe TBI (Glasgow score between 3 and 12 in the 24 first hours);
* At least 6 months following TBI;
* Complaint related to working memory in daily life (scale > 29 of questionnaire of complaint on working memory (WMQ), and established deficit of working memory by one of the following criteria:

  1. Index of working memory (IWM) of Wechsler Adult Intelligence Scale (WAIS-IV) < 85 or p < .05 between IWM and one of the WAIS-IV index;
  2. Less than 70% correct responses on Brown-Peterson tasks test in the verbal modality with an interfering task as mental calculation;
  3. Less than 89% correct responses on Brown-Peterson tasks test in the verbal modality with an interfering task of articulatory suppression;
  4. Less than 70% correct responses on Brown-Peterson tasks test in the visuospatial modality with an interfering motor task.
* Prior medical examination;
* Correct vision after visual acuity correction;
* Stable neurological or psychoactive treatment for at least 4 weeks, if applicable;
* Able to move to the center where rehabilitation will be performed;
* Covered by a health insurance;
* Signed consent of patient or of the guardian.

Exclusion Criteria:

* History of central nervous system disorder, or history of psychological disorder or substance abuse;
* Prior specific cognitive rehabilitation of working memory;
* Instrumental activities disabilities, cognitive disorder, behavioural disorders or major psychiatric disorder;
* Major anxio-depressive syndrome or present psychiatric disorder which can interfere with experimental procedure or measured variables;
* Pregnant or breastfeeding woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Proportions of simultaneous responders | 3 months after the first rehabilitation session
  A patient will be considered as a responder if he improves simultaneously on the Working Memory Questionnaire (WMQ) and the Brown-Peterson Task.
  Proportions will be calculated of patients simultaneously improving on the Working Memory Questionnaire (WMQ) and the Brown-Peterson Task:
  * increase of at least 12 points on WMQ scale,
  * at least 13% score improvement on the verbal or visuo-spatial Brown-Peterson Task.

SECONDARY OUTCOMES:
Working Memory Questionnaire during rehabilitation program | At baseline, 3 months, 6 months and 9 months
  The Working Memory Questionnaire (WMQ), an auto-questionnaire elaborated by the study team, will be used.
  The WMQ is a self-administered scale, addressing three dimensions of working memory: short-term storage, attention, and executive control.
  It is a self-assessment questionnaire comprising 30 questions scored on a five-point Likert scale, ranging from 0 ("no problem at all") to 4 ("very severe problem in everyday life"). The total score will be used.
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  Working memory span tasks
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  Verbal and visuospatial working memory.
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  n-back task
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  Brown-Peterson Visual.
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  reading span task.
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  Working Memory Index (WISC-IV).
Cognitive task of working memory | At baseline, 3 months, 6 months and 9 months
  divided attention task
Arithmetic resolution | At baseline, 3 months and 6 months
  Non-specific tasks involving working memory: arithmetic resolution ability by WAIS index
Non-targeted cognitive measurements | At baseline, 3 months and 6 months
  Executive functions will be assessed.
Non-targeted cognitive measurements | At baseline, 3 months and 6 months
  Long-term memory will be assessed.
Non-targeted cognitive measurements | At baseline, 3 months and 6 months
  The speed of treatment will be assessed.
Social functioning assessement | At baseline, 3 months, 6 months and 9 months
  Assessed by Manual for Sydney Psychosocial Reintegration Scale (SPRS)
Quality of life assessment | At baseline, 3 months, 6 months and 9 months
  Assessed by Qolibri scale
Quality of life assessment | At baseline, 3 months, 6 months and 9 months
  Assessed by EQ5D-5
Acceptability | At baseline, 3 months and 6 months
  Compliance of rehabilitation program: duration of training of speech-language pathologist and psychologist to the rehabilitation program.
Acceptability | At baseline, 3 months and 6 months
  Compliance of rehabilitation program: duration of session.
Acceptability | At baseline, 3 months and 6 months
  Compliance of rehabilitation program: patient's satisfaction of care (Client Satisfaction Questionnaire (CSQ-8)).
Acceptability | At baseline, 3 months and 6 months
  Compliance of rehabilitation program: presence during rehabilitation session of working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Vallat-Azouvi, PhD, Principal Investigator — Laboratoire LPN, EA2027-Université Paris 8, and Hôpital Raymond Poicaré-Antenne UEROS-UGECAMIDF; Philippe Azouvi, MD, PhD, Study Director — Service Médecine Physique et de Réadaptation, Hôpital Raymond Poicaré, 92380 Garches
Locations (1):
- Physical medicine and rehabilitation department, Raymond Poincaré Hospital, Garches, Hauts-de-seine, France

IPD SHARING:
Plan to Share IPD: No